CLINICAL TRIAL: NCT06572774
Title: An Integrated Community Clinic Model of Optimized Implementation Strategies to Increase Early Detection of Breast and Cervical Cancers in Kenya
Brief Title: Community Clinic Model to Improve Early Detection of Breast and Cervical Cancers in Kenya
Acronym: C3Link
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Implenomics (Other)
Collaborators: Kenya Medical Research Institute (Other); RTI International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Imp002
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Cervical Cancer
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: We are randomly assigning women to the three study arms. We are also requesting that the women select one caregiver for inclusion in the caregiver education sessions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- C3Link strategies (Experimental): Community liaison will host group education sessions and facilitate cervical and breast cancer screening
  Interventions: Behavioral: C3Link Strategies
- C3Link Plus Strategies (Experimental): In addition to group education sessions, the Community Liaison will offer women one-on-one education, counseling and navigation support to address barriers.
  Interventions: Behavioral: C3Link Strategies
- One-time education (Active Comparator): Participants will receive educational brochure on importance of breast and cervical cancer screening
  Interventions: Behavioral: C3Link Strategies

INTERVENTIONS:
Behavioral: C3Link Strategies — Education sessions and community liaison support to link to services

SUMMARY:
Kenya has a high incidence of breast and cervical cancers, and most women are diagnosed with late-stage disease. The investigators will conduct a study to assess the effectiveness and cost-effectiveness of strategies to increase the uptake of cancer screening and completion of recommended diagnostic and treatment services. The findings can be used to design optimal approaches and plan investments in infrastructure to scale up implementation of breast and cervical cancer screening.

DETAILED DESCRIPTION:
Kenya has a high incidence of breast and cervical cancers, and most women are diagnosed with late-stage disease. Implementing effective programs to screen and detect these cancers at an early stage could substantially decrease the high mortality. Kenya has been increasing access to cancer screening, but less than one-sixth of eligible women have ever received breast and cervical cancer screening.

The goal of the study is to assess the effectiveness and cost-effectiveness of multicomponent strategies to increase the uptake of breast and cervical cancer screening. A key gap that perpetuates the low screening rates in Kenya is the lack of community-clinic linkages. There is evidence that women are often unaware of the screening services offered in facilities, and, even among those who are aware, there is lack of motivation, anticipated or perceived stigma, and reduced self-efficacy to undergo screening. The investigators will conduct a pragmatic cluster randomized trial to evaluate the screening outcomes, including screening uptake, diagnostic test completion, and treatment initiation and implementation outcomes to support scale-up. The investigators will test two multicomponent packages of strategies: (1) Cancer Community-Clinic Linkage (C3Link) Core: Community health volunteer (CHV)-delivered group education for women and family members to increase screening uptake in the community setting and practice facilitation to improve the screening process and develop team-based care with CHV participation in the clinic setting; (2) C3Link Plus: C3Link Core strategies along with a sequential series of individual strategies that increase in intensity at 3-month intervals; women who remain unscreened will first receive one-on-one education; second, motivational interviewing; and, finally, navigation to address specific barriers.

The investigators will implement the study across 27 communities in Kenya to address the following three specific aims: Aim 1: Conduct a cluster randomized trial to assess short-term (intervention implementation phase) and longer-term impacts (maintenance phase) of the two packages of multicomponent strategies on breast and cervical cancer screening outcomes along the continuum of care compared to enhanced standard of care (communities receiving a messaging campaign only); Aim 2: Use a mixed-methods approach to assess and compare multilevel implementation outcomes of the package of strategies focusing on acceptability, feasibility, appropriateness, fidelity, and sustainability; Aim 3: Perform cost-effectiveness and return-on-investment analysis to support scale-up of an effective package of implementation strategies across Kenya and other sub-Saharan African countries. The Kenyan Ministry of Health can use the findings from this study to design optimal approaches and plan investments in screening infrastructure to scale up implementation of guideline recommendations. The lessons learned can be applied to other sub-Saharan African settings.

ELIGIBILITY:
Inclusion Criteria:

* Women will be eligible to participate if they are 30 to 55 years old, due to receive both breast and cervical cancer screening during the study intervention implementation phase based on Kenyan guideline recommendations, not experiencing breast or cervical cancer symptoms (will be referred for diagnostic testing with facilitation support from the study team), not pregnant, fluent in a study language (English,Kiswahili, Kamba, Kalenjin, and Kikuyu) and plan to remain in the community for at least 2 years

Exclusion Criteria:

-

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5400 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Breast and cervical cancer screening | 24 months
  The primary endpoint is the proportion who complete both recommended breast and cervical cancer screenings at 24 months

SECONDARY OUTCOMES:
Follow-up diagnostic procedure | 24 months
  Proportion who complete recommended follow-up supplemental or diagnostic procedures (within 3 months of receiving follow-up referral)
Initiation of cancer treatment | 24 months
  Proportion who initiative cancer treatment (within 3 months of diagnosis)

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health Facilities in Machakos, Nyeri and Nakuru, Machakos, Kenya